CLINICAL TRIAL: NCT04051567
Title: Low-dose Aspirin for Prevention of Adverse Pregnancy Outcomes in Twin Pregnancies--A Multicenter, Prospective, Open, Randomized, Controlled Clinical Trial
Brief Title: Low-dose Aspirin for Prevention of Adverse Pregnancy Outcomes in Twin Pregnancies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: Peking University Third Hospital (Other); Chongqing Medical Center for Women and Children (Other)
Responsible Party: Principal Investigator, Hongbo Qi, Professor, Ministry of Science and Technology of the People´s Republic of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: M2017047
Record Dates: First submitted 2019-07-09; First posted 2019-08-09 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Twin Pregnancy; Preeclampsia; Preterm Birth; Fetal Growth Restriction
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Fetal Growth Retardation | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LDA group (Experimental)
  Interventions: Drug: Aspirin 100mg
- NC group (No Intervention)

INTERVENTIONS:
Drug: Aspirin 100mg — In LDA group, patients were asked for taking 100mg aspirin per night;
  Arms: LDA group

SUMMARY:
Twin pregnancies are associated with increased risk of perinatal adverse outcomes , including preeclampsia , fetal growth restriction , preterm premature rupture of membranes and preterm birth. Low-dose aspirin was recommend by American College of Obstetricians and Gynecologists (ACOG) during pregnancy. In this trial, the investigators suppose that aspirin used in twin-pregnancies could improve adverse pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancy diagnosed by ultrasound and maternal age ranged from 18 to 55 years, Gestational age was less than 16w

Exclusion Criteria:

* Diagnosed fetal anomalies, history of cervical cerclage, contraindications of aspirin, pre-existing renal or liver diseases or abnormal functions, coagulation disorders, history of PE, preterm birth or FGR, chronic hypertension

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 425 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of preeclampsia, preterm birth, fetal growth restriction | after 30 weeks of gestional age

CONTACTS AND LOCATIONS:
Locations (1):
- Hongbo,Qi, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided